CLINICAL TRIAL: NCT05126225
Title: Buddhist Understanding and Reduction of Myanmar Experiences of HIV Stigma and Exclusion
Acronym: BURMESE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Chiangmai Rajabhat University (Unknown); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Weiti Chen, RN, CNM, PhD, FAAN, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB# 18-001769; R21TW011277 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hiv; Stigma, Social; Mindfulness
Keywords: stigma; Mindfulness; Myanmar
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Intervention Model Description: The intervention is modularized to have eight weekly sessions of 2-hour group discussions, led by a trained facilitator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protocol group (Experimental): The intervention is modularized to eight weekly sessions of 2-hour group discussions. The facilitator applies the principle of Cognitive Behavior Therapy and provides psychoeducation to promote the awareness and understanding of HIV stigma as well as training to help participants acquire alternative coping skills, such as relaxation techniques. In five sessions, participants are introduced to the general cognitive-behavioral model of HIV stigma and are encouraged to track their thoughts, feelings, and behavioral responses when encountering external stigma or adverse events. The participants further learn to differentiate helpful and non-helpful coping strategies and practice applying helpful coping skills to effectively reduce their HIV stigma. In the other three sessions, participants further discuss more specific stigma that intersects with HIV stigma, including stigma in healthcare settings, access to social support, and available resources on the society levels.
  Interventions: Behavioral: Stigma reduction

INTERVENTIONS:
Behavioral: Stigma reduction — The intervention is modularized to have eight weekly sessions of 2-hour group discussions, led by a trained facilitator. The facilitator applies the principle of CBT and provides psychoeducation to promote the awareness and understanding of HIV stigma as well as training to help participants acquire alternative coping skills, such as relaxation techniques.

SUMMARY:
This project aims to explore a multi-leveled conceptualization of the effects of HIV stigma on HIV care engagement in Myanmar by conducting a mixed-method study.

DETAILED DESCRIPTION:
This project is to explore how Myanmar People Living With HIV (PLWH) experience and manage HIV stigma as inspired by Buddhist teaching, and to adapt an evidence-based stigma-reduction intervention to tailor treatment for the unique needs of Myanmar People Living With HIV.

A stigma-reduction intervention will be adopted to the needs of Myanmar People Living With HIV with six focus groups.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-Positive
2. Care by Myanmar Positive Group/CMRU
3. Living in Myanmar/Thailand
4. can stay in the period of intervention

Exclusion Criteria:

1. Not HIV
2. Living outside of Myanmar/Thailand
3. Not care by MPG/CMRU
4. Cannot stay for the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Myanmar Positive Group, Yangon, Myanmar, Burma
- Chiangmai Rajabhat University, Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data upon request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The mixed methods study included interviews (n=32), focus groups (n=60) and a single arm interventional trial (n=19). The first part of the study consisted of interviews and focus groups from different stakeholders (PLWH, healthcare providers, family members, friends, etc.) which gathered data that was used to inform the intervention; outcomes were not collected from these participants. The second part of the study implemented the intervention in a single-arm pilot study with PLWH participants.
Groups:
- Interview Group: To explore how PLWH experience and interpret HIV stigma in Myanmar and then identify key sociocultural factors, and, in particular, key components of Buddhism, which may shape PLWH's experiences of stigma, we conducted in-depth interviews during Phase 1 of the study. The participants making up the interview group were used to inform the adaptation of an existing intervention for use in people living with HIV from Myanmar. Outcomes were not collected from participants who participated in the interviews since they did not receive the study intervention.
- Focus Group: After the initial adaption based on interviews, the first draft of the adapted intervention was presented to focus groups of Myanmar people living with HIV. A trained facilitator that matched the focus group members demographically led the discussions after the presentation of each module. All the discussion sessions were audiotaped. The focus group members completed a brief survey containing closed- and open-ended questions regarding the cultural appropriateness of various intervention components, including materials, metaphors, didactic methods, homework, and other content. Since the purpose of the feedback collected from focus groups was to judge the appropriateness, acceptability and feasibility of the adapted study intervention for use in the target population, outcomes were not collected from the focus group participants.
Period: Overall Study
Arm/Group | Protocol Group | Interview Group | Focus Group
Started | 19 | 32 | 60
Completed | 19 | 32 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Protocol Group: The protocol group was comprised of the participants who received the final, adapted study intervention over the course of 8 weeks.
  The intervention is modularized to eight weekly sessions of 2-hour group discussions. The facilitator applies the principle of Cognitive Behavior Therapy and provides psychoeducation to promote the awareness and understanding of HIV stigma as well as training to help participants acquire alternative coping skills, such as relaxation techniques. In five sessions, participants are introduced to the general cognitive-behavioral model of HIV stigma and are encouraged to track their thoughts, feelings, and behavioral responses when encountering external stigma or adverse events. The participants further learn to differentiate helpful and non-helpful coping strategies and practice applying helpful coping skills to effectively reduce their HIV stigma. In the other three sessions, participants further discuss more specific stigma that intersects with HIV stigma, including stigma in healthcare settings, access to social support, and available resources on the society levels.
  Stigma reduction: The intervention is modularized to have eight weekly sessions of 2-hour group discussions, led by a trained facilitator. The facilitator applies the principle of CBT and provides psychoeducation to promote the awareness and understanding of HIV stigma as well as training to help participants acquire alternative coping skills, such as relaxation techniques.
- Interview Group: Interviews were conducted during the first phase of the study. With the goal of culturally adapting an existing intervention for use among people living with HIV from Myanmar, in-depth interviews were conducted with people living with HIV from Myanmar to explore and identify Buddhist conceptualizations of HIV stigma. Participants in the interview group were not followed for outcomes or AEs.
- Focus Group: During the second step of the study, focus groups made up of Myanmar people living with HIV were presented the adapted intervention. Feasibility, acceptability, and appropriateness was assessed that informed the final version of the adapted study intervention for use in the target population. Participants in the focus group were not followed for outcomes or AEs.
- Total: Total of all reporting groups
Arm/Group | Protocol Group | Interview Group | Focus Group | Total
Number analyzed (Participants) | 19 | 32 | 60 | 111
Age, Continuous [Mean (Full Range); unit: years] | 35.4 [19 to 53] | 39 [18 to 49] | 39 [27 to 61] | 37.8 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 20 | 49
  Male | 10 | 12 | 40 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 32 | 60 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 19 | 32 | 60 | 111
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Stigma score [Mean (Standard Deviation); unit: score] — Perceived Stigma Scale (PSS). Each item measured using a 4-point Likert scale and the scale contains four factors: personalized stigma (18 items, subscore total 18-72), disclosure concerns (12 items, subscore total 12-48), negative self-image (9 items, subscore total 9-36), and concern with public attitudes about PLWH (12 items, subscore total 12-48). Each factor is scored separately. PSS score computed by summing 40 items, with a minimum total 40 and maximum score 160. Raw PSS scores were transformed into Stigma scores 1-4. Higher scores reflect higher levels of perceived stigma. Population: The baseline stigma score was not collected from the interview and focus group participants.
  score
    number analyzed (Participants) | 19 | 0 | 0 | 19
    (all) | 2.2358 (.56062) |  |  | 2.2358 (.56062)

OUTCOME MEASURES:

1. Primary Outcome: Change in Stigma Score From Baseline to End of Intervention in Protocol Group
Description: Perceived Stigma Scale (PSS). Each item is measured using a 4-point Likert scale and the scale contains four factors: personalized stigma (18 items, subscore total 18-72), disclosure concerns (12 items, subscore total 12-48), negative self-image (9 items, subscore total 9-36), and concern with public attitudes about people with HIV (12 items, subscore total 12-48). Each factor is scored separately, with total score is computed by summing all 40 items, with a minimum total PSS score of 40 and a maximum possible score of 160. Raw PSS scores were transformed into Stigma scores 1-4. Higher scores reflect higher levels of perceived stigma.
Time Frame: Baseline and 8 weeks
Population: Single-arm analysis was conducted in the protocol group.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Protocol group
Number analyzed (Participants) | 19
score
  Pre-test stigma score | 2.2358 (.56062)
  Post-test stigma score | 2.1760 (.69976)
Statistical Analysis 1: Comparison: Protocol group; Test type: Other — Single group; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [0.032 to 0.960], Standard Error of Mean 0.224

2. Secondary Outcome: Change in QOL Score From Baseline to End of Intervention in the Protocol Group
Description: Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is a 12-item questionnaire that was used as a proxy measure of QOL in the study. Total maximum score of CAMS-R is 48 and minimum score is 12. Raw CAMS-R scores were transformed into QOL scores 0-3. Higher scores reflect better QOL.
Time Frame: Baseline and 8 weeks
Population: Single-arm analysis was conducted in the protocol group.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Protocol group
Number analyzed (Participants) | 19
score
  Pre-test QOL score | 2.73 (0.82)
  Post-test QOL score | 2.68 (0.90)
Statistical Analysis 1: Comparison: Protocol group; Test type: Other — Single group; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.160 to 0.440], Standard Error of Mean 0.067

ADVERSE EVENTS:
Time Frame: AEs were collected weekly over a period of 8 weeks in the protocol group.
Description: Since the purpose of the first phase of the study was to adapt an existing intervention for use in the target population, adverse events were not collected from the participants in the interview and focus groups. Participants in the protocol group were assessed for adverse events over a span of 8 weeks while receiving the study intervention.
Arm/Group | Protocol Group
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
A small sample size limits the statistical power of a study, making it difficult to detect meaningful differences or relationships even if they exist. This can result in non-significant findings and wide confidence intervals, reducing confidence in the estimated effect size. Consequently, the results may not accurately represent the population or reflect the true effectiveness of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT05126225/Prot_SAP_000.pdf